CLINICAL TRIAL: NCT07217743
Title: Prospective, Single Center, Open-label Study Assessing Impact of Poly-L-lactic Acid on Adipogenesis in Patients on Glucagon-like Peptide-1 Agonists
Brief Title: Assess Impact of Poly-L-lactic Acid on GLP1 Subjects
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sculptra-Aesthetic-GLP1
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Laxity; Skin
Keywords: laxity; loose skin; glp1; abdominal laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: All subjects (15 GLP1 and 5 non GLP1) will receive three treatments, one month apart, of Sculptra Aesthetic to the abdomen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- GLP1 Patients (Active Comparator): 15 Participants who have been on a stable dose of GLP1 for at least 6 months will receive three treatments, one month apart, of Sculptra Aesthetic up to 16cc.
  Interventions: Device: Sculptra Aesthetic
- NON GLP1 Patients (Experimental): 5 participants who are GLP1 naive will receive three treatments, one month apart, of Sculptra Aesthetic up to 16cc.
  Interventions: Device: Sculptra Aesthetic

INTERVENTIONS:
Device: Sculptra Aesthetic — 15 GLP1 subjects treated with Sculptra to their abdomen for skin laxity will be compared to 5 non GLP1 subjects treated with Sculptra for skin laxity.

SUMMARY:
Clinical trial to evaluate treatments of double-dilute poly-L-lactic acid on abdominal skin laxity in GLP1 patients versus non GLP1 patients.

DETAILED DESCRIPTION:
20 patients total (15 GLP1 and 5 non-GLP1) will receive three treatments of double-dilute PLLA (Sculptra® Aesthetic; Galderma Laboratories; Fort Worth, TX) to the abdomen one month apart. Using a 22 G 2" cannula, up to 16cc of poly-L-lactic acid will be used per treatment. Patients will return for follow up visits at month 3 and month 9, where they will undergo standardized 2D photography and assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 25-65 years.
2. Fitzpatrick skin types I-IV.
3. Presence of mild to moderate skin laxity of abdomen, as determined by clinical investigators.
4. Stable weight for 3 months, with body mass index (BMI) of 27 or less.
5. Current treatment with a stable dose of GLP-1 agonist medication for at least the last 6 months, for 15 of the enrolled subjects. Remaining 5 subjects should not be taking or have a history of taking a GLP-1 agonist medication, and should not be planning to take a GLP-1 in the foreseeable future.
6. Must be willing to sign a photography release and ICF, and complete the entire course of the study.
7. Subjects in good general health based on investigator's judgment and medical history.
8. Negative urine pregnancy test result at the time of study entry (if applicable).
9. Subjects of childbearing potential must agree to use an effective method of birth control during the entire course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment.

   1. Acceptable forms of birth control are: oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device/coil, double-barrier methods (e.g., sponge, spermicide, or condoms). Abstinence and/or vasectomized partner must agree to a second acceptable method of birth control (double-barrier) should the subject become sexually active.
   2. A female is considered of non-childbearing potential if she is: postmenopausal (no menses for at least 12 months), without a uterus (hysterectomy) and/or both ovaries (oophorectomy), or bilateral tubal ligation.

Exclusion Criteria:

1. The presence of severe abdominal skin laxity as determined by clinical investigators.
2. Still actively losing weight.
3. Pregnancy or planned pregnancy during the study or currently breastfeeding.
4. Any uncontrolled systemic disease.
5. History of autoimmune connective tissue disease.
6. Current use of immunosuppressive medication.
7. Significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
8. Active dermatitis or active infection in the proposed treatment area.
9. Mesotherapy; dermal fillers, biostimulator injectables; radiofrequency device treatments; microfocused ultrasound device treatments; laser and light-based device treatments; microneedling; cryolipolysis; high intensity focused electromagnetic energy device treatment; or surgery during the 12-month period before study treatment.
10. Any investigational treatment for skin quality of the abdomen during the 12-month period before the study treatment
11. Creams/cosmeceuticals and/or home therapies for the prevention or treatment of skin quality in the treatment area during the 1-month period before study treatment
12. Subjects with scarring in the treatment areas, including laparoscopic or abdominal surgery scars, which in the opinion of the investigator could impact results. Subjects with a history of keloids will be excluded.
13. Subjects who spray tanned or used sunless tanners in the treatment areas 1-month prior to study treatment.
14. History of bleeding disorder, concomitant use of anticoagulants, history of connective tissue disease (e.g., lupus, scleroderma), history of Bell's Palsy, epilepsy, smoking, and/or current pregnancy or breastfeeding .
15. Inability to ambulate following the procedure.
16. History of lidocaine and/or epinephrine sensitivity deemed by the investigator to preclude subject from enrolling into study.
17. Individuals with known allergies or sensitivities to any of the ingredients of any topical or injectable products being used in this study.
18. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female at birth
Enrollment: 20 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Physical Global Aesthetic Improvement Scale | Month 3 and Month 9
  Assess improvement of Abdominal skin laxity:
  Much Improved 2 Improved 1 No Change 0 Worse -1 Much Worse -2

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale | Month 3 and Month 9
  Assess improvement of Abdominal skin laxity:
  Much Improved 2 Improved 1 No Change 0 Worse -1 Much Worse -2

CONTACTS AND LOCATIONS:
Locations (1):
- West Dermatology Research Center, San Diego, California, United States